CLINICAL TRIAL: NCT00421538
Title: Contention Alone Versus Anticoagulation for Symptomatic Calf Vein Thrombosis Diagnosed by Ultrasonography
Brief Title: Randomized Controlled Trial of Anticoagulation vs. Placebo for a First Symptomatic Isolated Distal Deep-vein Thrombosis (IDDVT)
Acronym: CACTUS-PTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss National Science Foundation (Other); Ministry of Health, France (Other Government); Lady Davis Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marc Righini, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3200B0-105991; CACTUS-PTS Trial; NCT00539058 (obsolete NCT alias)
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Distal (Calf) Deep-vein Thrombosis
Keywords: Deep vein Thrombosis; Calf vein thrombosis; Low-molecular weight heparin; Placebo; Elastic contention; Compression Ultrasonography
MeSH Terms: conditions — Venous Thrombosis | interventions — Nadroparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMWH (Active Comparator): Therapeutic dose of Nadroparin
  Interventions: Drug: nadroparine calcium
- Placebo (Placebo Comparator): Injectable placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: nadroparine calcium — Once-daily injection of 171 U/Kg/day of nadroparine calcium for 6 weeks.
  Arms: LMWH
Drug: Placebo — Once-daily injectable placebo (sterilized NaCL 0.9%) for 6 weeks
  Arms: Placebo

SUMMARY:
CACTUS-PTS is a randomized, placebo-controlled, double-blind study which aims primarily to determine the effectiveness of a 6 week course of therapeutic-dose LMWH (nadroparine) injections vs. placebo in patients with a first symptomatic isolated distal (calf) deep-vein thrombosis (IDDVT), as measured by rate of proximal DVT and symptomatic PE at 6 weeks. Additionally, the study aims to determine if the 6 week course of treatment with therapeutic-dose LMWH (nadroparine) injections, compared to placebo, decreases the frequency of post-thrombotic syndrome (PTS) at 1 year.

DETAILED DESCRIPTION:
The CACTUS-PTS study will compare anticoagulant treatment for 6 weeks versus placebo in acute, symptomatic distal DVT. Patients will be randomized to receive either a six-week period of LMWH at therapeutic dosage or a six-week period of placebo. All patients will be treated with elastic compression stockings and followed-up with a standardized ultrasonography protocol. Strict ultrasonographic diagnostic criteria for distal DVT have been defined. Control compression ultrasonography will be performed between days 3 and 7 and at six weeks after inclusion. The primary outcome will be a composite of the proportion of patients with extension of the thrombus to the proximal veins (detected by the programmed ultrasound examinations or by an ultrasound performed because of recurrent symptoms) or symptomatic PE in both arms of the study during the 6-weeks study period. Patients with such an outcome will be anticoagulated as currently admitted in presence of a proximal DVT. Secondary outcomes will be the individual components of the composite endpoint (distal DVT extension to proximal veins; symptomatic PE), major bleeding, serious adverse events and death reported at 6 weeks and 90 days. To answer the research question of the PTS add-on study, patients will self-assess and be assessed for PTS by a clinician using the Villalta scale, 1 year following their enrolment into the trial. In addition, patients will complete a Quality of Life (QOL) questionnaire. The QOL questionnaire will be comprised of both the VEINES-QOL and SF-36. The primary outcome is the rate of PTS, with secondary outcomes of QOL scores and PTS severity.

ELIGIBILITY:
Inclusion Criteria:

* All outpatients with an acute, symptomatic, distal DVT will be included in the study, provided they correspond to the following diagnostic and exclusion criteria, and they have signed an informed consent form.

Exclusion Criteria:

* Age less than 18 years
* Previously objectively diagnosed DVT or PE
* Distal DVT involving the tibioperoneal trunk (i.e. calf trifurcation)
* Clinically suspected pulmonary embolism
* Active cancer, receiving cancer treatment or cancer considered cured for <6 months
* Ipsilateral or contralateral proximal DVT
* Indication for long-term anticoagulation (e.g. atrial fibrillation, mechanical heart valve...)
* Pregnancy
* Thrombocytopenia (platelet count < 100 g/l)
* Impaired renal function (serum creatinine > 180 micromol/l or clearance to creatinine less than 30 ml/min)
* Known hypersensitivity to heparin
* Presence of an active bleeding or a pathology susceptible of bleeding in presence of anticoagulation (gastric ulcer, cerebral malignant disease...)
* Treatment with daily NSAIDs (aspirin ≤160 mg/day permitted)
* Body weight >115 kg or <40 kg
* Treatment with therapeutic doses of anticoagulants for >2 days, corresponding to: 2 injections of LMWH if once daily therapeutic LMWH used; 3 injections of LMWH if twice-daily therapeutic LMWH used; 1 dose of oral vitamin K antagonist (e.g. warfarin)
* Ongoing requirement for prophylactic dose thromboprophylaxis (e.g. acute post-op patient receiving thromboprophylaxis)
* Enrolled in another clinical trial within previous 30 days
* Inability or refusal to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Composite of rate of extension of distal DVT to proximal deep veins (includes ipsilateral extension or new contralateral proximal DVT) or symptomatic PE at 6 weeks | 6 weeks
Rate of post-thrombotic syndrome (PTS) | 1 year
  Rate of post-thrombotic syndrome (PTS) diagnosed using the Villalta scale.

SECONDARY OUTCOMES:
Individual components of the composite endpoint: distal DVT extension to proximal veins at 6 weeks and 90 days; PE at 6 weeks and 90 days | 6 weeks and 3 months
Major bleeding at 6 weeks and 90 days | 6 weeks and 3 months
Death at 6 weeks and 90 days | 6 weeks and 3 months
Serious adverse events at 6 weeks and 90 days | 6 weeks and 3 months
Generic and venous disease-specific Quality of Life scores | 1 year
PTS severity category | 1 year
  Can either be mild, intermediate, severe

CONTACTS AND LOCATIONS:
Overall Officials: Marc Righini, MD, Principal Investigator — University Hospital, Geneva; Isabelle Quéré, MD, Principal Investigator — Montpellier University Hospital; Susan Kahn, MD, Principal Investigator — Jewish General Hospital; Marc Carrier, MD, Principal Investigator — Ottawa Hospital
Locations (7):
- Canada (5):
  - Hamilton General Hospital, Hamilton, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Montpellier University Hospital, Montpellier, Languedoc, France
- University Hospital of Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Righini M, Robert-Ebadi H, Glauser F, Blondon M, Ouvry P, Diamand JM, Tissot A, Frappe P, Quere I, Kahn SR, Galanaud JP, Le Gal G. Effect of anticoagulant treatment on pain in distal deep vein thrombosis: an ancillary analysis from the cactus trial. J Thromb Haemost. 2019 Mar;17(3):507-510. doi: 10.1111/jth.14387. Epub 2019 Feb 3. PMID 30656824
- [Derived] Righini M, Galanaud JP, Guenneguez H, Brisot D, Diard A, Faisse P, Barrellier MT, Hamel-Desnos C, Jurus C, Pichot O, Martin M, Mazzolai L, Choquenet C, Accassat S, Robert-Ebadi H, Carrier M, Le Gal G, Mermilllod B, Laroche JP, Bounameaux H, Perrier A, Kahn SR, Quere I. Anticoagulant therapy for symptomatic calf deep vein thrombosis (CACTUS): a randomised, double-blind, placebo-controlled trial. Lancet Haematol. 2016 Dec;3(12):e556-e562. doi: 10.1016/S2352-3026(16)30131-4. Epub 2016 Nov 8. PMID 27836513
- [Derived] Guanella R, Righini M. Serial limited versus single complete compression ultrasonography for the diagnosis of lower extremity deep vein thrombosis. Semin Respir Crit Care Med. 2012 Apr;33(2):144-50. doi: 10.1055/s-0032-1311793. Epub 2012 May 30. PMID 22648486